CLINICAL TRIAL: NCT05362318
Title: Motivating Smoking Cessation and Relapse Prevention Among Lung Cancer Patients: Helping and Empowering pAtients for Living a Life Smoke-free (Project HEALS)
Brief Title: Project HEALS (Helping and Empowering pAtients for Living a Life Smoke-free
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-21108
Record Dates: First submitted 2022-04-29; First posted 2022-05-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Smoking; Tobacco Use; Lung Cancer
MeSH Terms: conditions — Smoking; Tobacco Use; Lung Neoplasms | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Usual Care (Active Comparator): Participants will receive brief advice to quit, an offer of enrollment to the Florida Tobacco Quitline, and a 12 week supply of nicotine replacement therapy (nicotine patches and lozenges).
  Interventions: Drug: Nicotine patch and lozenges; Behavioral: Florida Tobacco Quitline
- Group 2: Usual Care + Motivation and Problem Solving + Relapse Prevention (Experimental): Participants will receive brief advice to quit, an offer of enrollment to the Florida Tobacco Quitline, and a 12 week supply of nicotine replacement therapy (nicotine patches and lozenges), 6 telephone counseling sessions over 6 months, and access to a web based video.
  Interventions: Drug: Nicotine patch and lozenges; Behavioral: Telephone counseling sessions; Behavioral: Access to a web-based video; Behavioral: Florida Tobacco Quitline

INTERVENTIONS:
Drug: Nicotine patch and lozenges — Participants will receive nicotine patch and lozenges. The regimen will be based on the participant's self-reported smoking rate. At the time of enrollment, a research staff member will determine the proper dose. Participants who smoke >10 cigarettes/day will receive 8 weeks of 21 mg. patches, 2 weeks of 14 mg. patches, 2 weeks of 7 mg. patches, and 12 weeks of 2 mg. lozenges. Those who smoke <10 cigarettes/day will receive 8 weeks of 14 mg. patches, 4 weeks of 7 mg patches, and 12 weeks of 2 mg. lozenges
Behavioral: Telephone counseling sessions — Participants will be offered 6 Motivation and Problem Solving (MAPS)-based counseling sessions by phone over a 6-month period.
  Arms: Group 2: Usual Care + Motivation and Problem Solving + Relapse Prevention
Behavioral: Access to a web-based video — Participants will be given web-based access to the relapse prevention video "Surviving Smokefree".
  Arms: Group 2: Usual Care + Motivation and Problem Solving + Relapse Prevention
Behavioral: Florida Tobacco Quitline — Participants will receive an offer of enrollment to the Florida Tobacco Quitline which enables participant to speak with a Quit Coach who will assess nicotine addiction and help create a quit plan.

SUMMARY:
The purpose of the study is to pilot test a multi-modal smoking cessation and relapse prevention intervention with the lung cancer patient population and to obtain preliminary data on its feasibility.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Smoked at least 100 cigarettes in lifetime
* Current smoking (defined as self-report of any smoking, even a puff, in the past 30 days)
* Diagnosis of lung cancer
* Able to read and write English
* Not currently enrolled in a smoking cessation program
* Has a working telephone
* Has a valid home address

Exclusion Criteria:

* Current use of tobacco cessation medications
* Another household member enrolled in this study
* Contraindication of nicotine patch, unless under the supervision of a physician as advised by project staff
* Moffitt clinical trial participant at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who meet inclusion criteria | Baseline
  Percentage of participants who meet inclusion criteria
Percentage of participants who agree to participate in the study | Baseline
  Percentage of participants who agree to participate in the study
Percentage of participants completing baseline assessment | Baseline
  Percentage of participants completing baseline assessment
Percentage of participants completing the 3 month follow-up assessments | at 3 months
  Percentage of participants completing the 3 month follow-up assessments
Percentage of participants completing the 6 month follow-up assessments | at 6 months
  Percentage of participants completing the 6 month follow-up assessments
Treatment satisfaction - Acceptability | at 6 months
  Mean scores of the Client Satisfaction Questionnaire (SCQ-8) will be used for this measure. The CSQ-8 comprises 8 items for the assessment of treatment satisfaction using a scale from 8 to 32, with higher scores indicating greater satisfaction.
Completion rate of MAPS calls for UC+MAPS+RP participants - Demand | at 6 months
  Percentage of MAPS calls completed for UC+MAPS+RP participants
Percentage of UC+MAPS+RP participants who viewed the web-based video -Demand | at 3 months
  Percentage of UC+MAPS+RP participants who viewed the web based video
Percentage of UC+MAPS+RP participants who viewed the web-based video -Demand | at 6 months
  Percentage of UC+MAPS+RP participants who viewed the web based video

CONTACTS AND LOCATIONS:
Overall Officials: Vani N Simmons, PhD, Principal Investigator — Moffitt Cancer Center; Jennifer I Vidrine, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided